CLINICAL TRIAL: NCT02743455
Title: A Phase I, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of MVA-BN Yellow Fever Vaccine With and Without Montanide ISA 720 Adjuvant in 18-45 Year Old Healthy Adults
Brief Title: A Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of MVA-BN Yellow Fever Vaccine With and Without Montanide ISA-720 Adjuvant in 18-45 Year Old Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0107; HHSN272201300020I
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2019-02-01

CONDITIONS: Yellow Fever; Yellow Fever Immunisation
Keywords: Fever; Immunogenicity; MVA-BN; Reactogenicity; Vaccine; Yellow
MeSH Terms: conditions — Yellow Fever; Fever | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Active Comparator): Subjects will receive 1.0x10^8 TCID50 of MVA-BN as two doses subcutaneously on Day 1 and Day 29. N=15
  Interventions: Biological: MVA Smallpox Vaccine
- Group 2 (Experimental): Subjects will receive 1.0x10^8 TCID50 of MVA-BN-YF as two doses intramuscularly on Day 1 and Day 29. N=15
  Interventions: Biological: MVA-BN Yellow Fever Vaccine
- Group 3 (Experimental): Subjects will receive 1.0x10^8 TCID50 of MVA-BN-YF + ISA 720 as two doses intramuscularly on Day 1 and Day 29. N=15
  Interventions: Drug: ISA-720; Biological: MVA-BN Yellow Fever Vaccine
- Group 4 (Experimental): Subjects will receive 1.0x10^8 TCID50 of MVA-BN-YF + ISA 720 as a single dose intramuscularly on Day 1 and matching placebo on Day 29. N=15
  Interventions: Drug: ISA-720; Biological: MVA-BN Yellow Fever Vaccine; Other: Placebo
- Group 5 (Active Comparator): Subjects will receive = / > 4.74 log10 PFU of YF-Vax as a single dose subcutaneously on Day 1 and matching placebo on Day 29. N=15
  Interventions: Other: Placebo; Biological: YF Vax 17D Strain
- Group 6 (Experimental): Subjects with prior receipt of MVA-BN will receive 1.0x10^8 TCID50 of MVA-BN-YF as two doses intramuscularly on Day 1 and Day 29. N=15
  Interventions: Biological: MVA-BN Yellow Fever Vaccine

INTERVENTIONS:
Drug: ISA-720 — The vaccine adjuvant ISA 720 will be used with Modified Vaccinia Ankara-Bavarian Nordic-Yellow Fever (MVA-BN-YF) as vaccine adjuvant with a depot effect. This comprises slow release of antigen at the injection site, protection of antigen against degradation and strong stimulation of the immune response.
  Arms: Group 3; Group 4
Biological: MVA Smallpox Vaccine — Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine (MVA BN(R)) is a purified live vaccine will be used as an active comparator.
  Arms: Group 1
Biological: MVA-BN Yellow Fever Vaccine — Modified Vaccinia Ankara-Bavarian Nordic-Yellow Fever (MVA-BN-YF) clinical trial material is manufactured in CEF cells derived from Specific Pathogen Free (SPF) eggs in a bioreactor culture using serum free medium.
  Arms: Group 2; Group 3; Group 4; Group 6
Other: Placebo — 0.9% Sodium Chloride Injection, USP is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection.
  Arms: Group 4
Other: Placebo — 0.9% Sodium Chloride Injection, USP is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection.
  Arms: Group 5
Biological: YF Vax 17D Strain — Yellow Fever Vaccine (YF-VAX) is a vaccine prepared by culturing the 17D-204 strain of yellow fever virus in living avian leucosis virus-free (ALV-free) chicken embryos. Will be used as an active comparator.
  Arms: Group 5

SUMMARY:
This study is a multi-center, double-blind, placebo-controlled, Phase I study to evaluate the safety, reactogenicity, tolerability, and immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic-Yellow Fever (MVA-BN-YF) in Flavivirus-naive healthy male and non-pregnant female adult subjects. There are six dose groups in this study. Subjects who have never received a licensed or investigational smallpox vaccine will be randomized to Groups 1-5 and vaccine administration and follow-up will be conducted in a double-blinded fashion. Subjects who have previously received two, 1 x 10^8 TCID50 doses of Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) between 19 and 45 days apart by s ubcutaneous (SC) or intramuscular (IM) routes will be enrolled in Group 6 and will be dosed open-label. Since this is a first in human, phase I study, a sentinel cohort will be utilized. The first two subjects (1st sentinel group) one at each clinical site will be randomized to Group 2 or 3 and vaccinated with MVA-BN-YF with or without Montanide ISA 720 adjuvant (ISA 720). Subjects and study personnel will be blinded as to whether ISA 720 was administered. The primary objectives are the: 1) assessment of the safety, tolerability, and reactogenicity of MVA-BN-YF vaccine administered with or without ISA 720; 2) comparison of the safety, tolerability, and reactogenicity of MVA-BN-YF vaccine administered with or without ISA 720 with Yellow Fever Vaccine (YF-VAX) and MVA-BN.

DETAILED DESCRIPTION:
This study is a multi-center, double-blind, placebo-controlled, Phase I study to evaluate the safety, reactogenicity, tolerability, and immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic-Yellow Fever (MVA-BN-YF) in Flavivirus-naive healthy male and non-pregnant female adult subjects. There are six dose groups in this study. Subjects who have never received a licensed or investigational smallpox vaccine will be randomized to Groups 1-5 and vaccine administration and follow-up will be conducted in a double-blinded fashion. Subjects who have previously received two, 1 x 10^8 TCID50 doses of Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) between 19 and 45 days apart by subcutaneous (SC) or intramuscular (IM) routes will be enrolled in Group 6 and will be dosed open-label. Since this is a first in human, phase I study, a sentinel cohort will be utilized. The first two subjects (1st sentinel group) one at each clinical site will be randomized to Group 2 or 3 and vaccinated with MVA-BN-YF with or without Montanide ISA 720 adjuvant (ISA 720). Subjects and study personnel will be blinded as to whether ISA 720 was administered. Subjects will be monitored for safety for one day, and if no pre-defined halting rule is met then two additional subjects (2nd sentinel group) one at each clinical site will be assigned to the group the previous subject was not assigned to. These subjects will be vaccinated and monitored as above. A total of 4 sentinel subjects will be vaccinated. The primary objectives are the: 1) assessment of the safety, tolerability, and reactogenicity of MVA-BN-YF vaccine administered with or without ISA 720; 2) comparison of the safety, tolerability, and reactogenicity of MVA-BN-YF vaccine administered with or without ISA 720 with Yellow Fever Vaccine (YF-VAX) and MVA-BN. The secondary objectives are the: 1) assessment of the immunogenicity against the MVA-BN backbone and Yellow Fever Virus (YF) antigen insert of MVA-BN-YF with and without ISA 720 as assessed by kinetics of the immune responses, seroconversion rates, and peak Geometric Mean Titer (GMT); 2) assessment of the impact of previous MVA-BN vaccination on peak immune responses to YF antigen in MVA-BN-YF; 3) comparison of the peak immunogenicity against YF antigen of 1 or 2 doses of MVA-BN-YF with or without ISA 720 with YF-VAX; 4) comparison of the peak immunogenicity against the MVA-BN backbone of 1 or 2 doses of MVA-BN-YF with or without ISA 720 with MVA-BN; 5) assessment of durability of immune response to YF antigen and MVA-BN at 6 months after 2nd vaccination or placebo administration.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male or female at least 18 to < / = 45 years old at the time of screening.
2. Must be able to read and provide written consent and complete the Informed Consent.
3. Must have a body mass index (BMI) > / = 18.5 and < 35.0 kg/m^2.
4. Must be in good health on the basis of physical examination, vital signs*, medical history, safety laboratories, and the investigator's clinical judgment. *Safety laboratory normal ranges will be those used by the reference clinical lab. Protocol-specific criteria for individual subjects are listed in criteria #6

   * The clinical laboratory evaluations that will be graded as laboratory Adverse Events (AEs) and be considered for the Study or Individual Halting Rules are those which are included in the laboratory toxicity grading scales.
   * Vital signs must be in normal ranges. If a subject has elevated systolic or diastolic blood pressure, subject may rest for 10 minutes in a quiet room and then the blood pressure may be retaken once.
5. For Group 6: subjects must have documented previous vaccination with MVA-BN*. *In order to be enrolled, a subject has to have received two 1x10^8 TCID50 doses of MVA-BN 19-45 days apart subcutaneous (SC) or intramuscular (IM) as part of participation in DMID vaccine trials 11-0021 or 09-0002. First dose must have been administered no earlier than 2010.
6. Must have acceptable* laboratory criteria within 28 days before enrollment.

   *Acceptable lab parameters include:
   * Hemoglobin: women: > 11.0 g/dL; men > 12.5 g/dL
   * White blood cell count: > 3,700 cells/mm^3 but < 11,000 cells/mm^3
   * Platelets: > 125,000 but < 375,000 per mm^3
   * Urine dipstick (clean urine sample): protein < 1+, glucose negative
   * Alanine aminotransferase and aspartate aminotransferase (ALT, AST) < 1.25 x institutional upper limit of normal
   * Blood urea nitrogen (BUN) < / = 1 x institutional upper limit of normal
   * Total bilirubin < 1.25x institutional upper limit of normal.
   * Serum creatinine < / = 1 x institutional upper limit of normal
   * If laboratory screening tests are out of range, repeat of screening tests is permitted once, provided there is an alternative explanation for the out of range value.
7. Women of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy tests prior to each vaccination.
8. Women of childbearing potential must have an acceptable method of contraception* from 28 days prior to the 1st vaccination until at least 60 days after the 2nd vaccination.

   *Acceptable methods of contraception include the following:

   -Prescription oral contraceptives, contraceptive injections, intrauterine device (IUD), implants, vaginal ring, double-barrier method, contraceptive patch, male partner sterilization, abstinence (defined as refraining from heterosexual intercourse during participation in the study [from 28 days before the first vaccination until at least 60 days after the last vaccination]). Women of non-childbearing potential, defined as postmenopausal (any age with amenorrhea for = / > 12 months without other known or suspected cause for amenorrhea, or surgically sterile (hysterectomy, bilateral tubal ligation, obilateral oophorectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure), are not required to use the birth control methods.
9. Female subjects must agree to not donate eggs (ova, oocytes) from the start of screening onwards until at least 60 days after the last vaccination.
10. Male subjects who have not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use an acceptable measure of birth control* from 28 days prior to 1st vaccination until at least 60 days after the last vaccination.

    *Acceptable methods of birth control include the following:
    * Abstinence (defined as refraining from heterosexual intercourse with a female partner of childbearing potential during participation in the study [from 28 days before the first vaccination until at least 60 days after the last vaccination].
    * A double-barrier method of birth control, such as condom with spermicidal foam/gel/film/cream/suppository and partner with occlusive cap (diaphragm, cervical/vault caps).
    * In case the female partner is using an acceptable method of birth control (see Inclusion Criterion #8), a single-barrier method of birth control for the male subject is acceptable.
11. Male subjects must agree to not donate sperm from the start of screening onwards until at least 60 days after the last vaccination.
12. Must be available and willing to participate for the duration of the study visits and follow-up.
13. Must have a means to be contacted by telephone.

Exclusion Criteria:

1. Was ever vaccinated with a licensed or investigational YF vaccine or was diagnosed with YF infection or disease*.

   *Includes YF-VAX, Stamaril, or Bio-Manguinhos yellow fever vaccine. Subject's verbal history will suffice.
2. Was ever vaccinated with a licensed or investigational Flavivirus vaccine*.

   *Including Japanese encephalitis virus (JEV) vaccine or an investigational Flavivirus vaccine including dengue virus (DENV) or West Nile virus vaccine, or has been diagnosed with an illness caused by a Flavivirus including DENV, West Nile virus (WNV), JEV, St. Louis encephalitis, or tick-borne encephalitis virus (TBEV). Subject's verbal history will suffice.
3. Positive serology for HIV, Hepatitis C virus, or Hepatitis B surface antigen.
4. Positive serology to Dengue, Yellow Fever, or West Nile virus.
5. Plans to travel to a Yellow-Fever endemic area during the course of the study* or travel to a Yellow-Fever endemic area within 30 days of screening.

   *Subjects who have a recent travel to a Yellow Fever endemic area may screen if they have returned to the U.S. 30 or more days prior to the screening visit. Refer to the CDC Yellow Fever map for countries/regions at risk for Yellow Fever virus infection. http://www.cdc.gov/yellowfever/maps/
6. Was ever vaccinated with a licensed or investigational smallpox vaccine* with the exception of subjects in Group 6.

   *Includes Dryvax, Acam2000, LC 16 m8, MVA-based vaccine candidate or licensed vaccines, and Imvamune or Imvanex.

   -EXCEPTION: Group 6 should have had two 1 x 10^8 TCID 50 doses of MVA-BN 19-45 days apart SC or IM as part of participation in DMID vaccine trials 11-0021 or 09-0002. First dose must have been administered no earlier than 2010.
7. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products*.

   *Including egg products, aminoglycosides, gelatin, sorbitol, tris (hydroxymethyl)-amino methane (THAM), or any of the constituents of the study vaccines.
8. Has severe allergy or anaphylaxis to latex*.

   *Participants in Group 6 will not be exposed to latex and so may have history of severe allergy or anaphylaxis to latex.
9. Has an acute illness or temperature > / = 38.0 degrees Celsius on Day 1 or Day 29*.

   *Subjects with fever or acute illness on the Day of vaccination may be re-assessed and enrolled if healthy or only minor residual symptoms remain within 3 days.
10. Female subjects who are pregnant or breast-feeding, or planning to become pregnant while enrolled in the study.
11. Has history of chronic or acute severe neurologic condition*.

    *Including history of seizure disorder or epilepsy, history of Guillain-Barre syndrome, Bell's palsy, meningitis, or disease with any focal neurologic deficits.
12. Has history of thymus disorder including myasthenia gravis, thymoma or prior thymectomy.
13. Has history of autoimmune disease, or clinically significant cardiac, pulmonary, hepatic, rheumatologic, or renal disease by history, physical examination, and/or laboratory studies*.

    *Includes the conditions and diagnoses defined as AESI.
14. Has history of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure*.

    *Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
15. Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy*.

    *Anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) are allowed.
16. Is post-organ and/or stem cell transplant whether or not on chronic immunosuppressive therapy.
17. Had major surgery (per the investigator's judgment) within the 4 weeks prior to study entry or planned major surgery during the course of the study.
18. Has personal history of recurring migraines (every 6 months or more often) or on prescription medication for treatment of recurring headaches or migraines.
19. Has history of cardiac disease*.

    *Myocarditis, pericarditis, cardiomyopathy, transient ischemic attack or stroke, myocardial infarction, angina, coronary artery disease, congestive heart failure, clinically significant arrhythmia. Includes any arrhythmia requiring medication, treatment, or clinical follow-up.
20. Has electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myocarditis/pericarditis*.

    *Including any of the following:
    * Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS = / > 120 ms, PR interval > 219 ms, any second-or third-degree atrioventricular block, or prolongation of the QT interval corrected according to Bazett's formula [QTcB] [> 450 ms]).
    * Significant repolarization (ST-segment or T-wave) abnormality.
    * Significant atrial or ventricular arrhythmia; frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, 2 premature ventricular contractions in a row).
    * ST-elevation consistent with ischemia or evidence of past or evolving myocardial infarction.
21. Has history of diabetes mellitus type 1 or type 2, including cases controlled with diet alone.

    -Note: history of isolated gestational diabetes is not an exclusion criterion.
22. Has history of thyroidectomy, or thyroid disease requiring medication during the last 12 months.
23. Has history of hypertension even if medically controlled.

    -Note: Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.
24. Received live attenuated vaccines from 30 days before Day 1 until 30 days after the 2nd vaccination.
25. Received killed or inactivated vaccines from 14 days before Day 1 until 14 days after the 2nd vaccination.
26. Received experimental therapeutic agents within 3 months prior to the first study vaccination or plans to receive any experimental therapeutic agents during the course of the study.
27. Is currently participating or plans to participate in another clinical study which would involve receipt of the following*:

    *An investigational product, blood drawing, or an invasive medical procedure that would require administration of anesthetics or intravenous dyes or removal of tissue during the study.

    -Includes endoscopy, bronchoscopy, or administration of IV contrast.
28. Received blood products or immunoglobulin in the 3 months before study entry or planned use during the course of the study.
29. Donated a unit of blood within 8 weeks before Day 1 or plans to donate blood during the course of the study.
30. Has major psychiatric illness during the past 12 months that in the opinion of the investigator would preclude participation.
31. Has current alcohol use or current or past abuse of recreational or narcotic drugs by history as judged by the investigator to potentially interfere with study adherence.
32. Has a history of chronic urticaria (recurrent hives).
33. Has tattoos, scars, or other marks on both deltoid areas which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
34. Is a study site employee* or staff who are paid entirely or partially by/through the OCRR contract for the trial, or staff who are supervised by the PI or Sub-Investigators.

    *Including the Principal Investigator (PI), sub-Investigators listed in Form FDA 1572 or Investigator of Record Form.
35. In the opinion of the investigator cannot communicate reliably, is unlikely to adhere to the requirements of the study, or has any condition which would limit the subject's ability to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Comparison of Grade 3 local, systemic or laboratory toxicities, continuous Grade 2 or greater local reactogenicity | Day 1 through Day 8
Comparison of Grade 3 local, systemic or laboratory toxicities, continuous Grade 2 or greater local reactogenicity | Day 29 through Day 36
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 1 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 2 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 3 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 4 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 5 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination in Group 6 | Day 1 through Day 394
Number of adverse events of special interest (AESIs) considered related to study vaccination overall | Day 1 through Day 394
Number of related adverse events of special interest (AESIs) | Day 1 through Day 394
Number of related serious adverse events (SAEs) | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 1 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 2 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 3 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 4 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 5 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination in Group 6 | Day 1 through Day 394
Number of serious adverse events (SAEs) considered related to study vaccination overall | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 1 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 2 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 3 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 4 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 5 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition in Group 6 | Day 1 through Day 394
Number of subjects with new onset of a chronic medical condition overall | Day 1 through Day 394
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 1 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 2 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 3 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 4 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 5 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) in Group 6 | Day 1 through Day 57
Number of subjects with unsolicited vaccine-related adverse events (AEs) overall | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 1 | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 2 | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 3 | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 4 | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 5 | Day 1 through Day 57
Number of vaccine-related laboratory adverse events (AEs) in Group 6 | Day 1 through Day 57
Number of withdrawals or discontinuation of vaccinations due to any reason | Day 1 through Day 394
Occurrence of solicited injection site reactogenicity events in Group 1 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 1 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events in Group 2 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 2 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events in Group 3 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 3 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events in Group 4 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 4 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events in Group 5 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 5 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events in Group 6 | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events in Group 6 | Day 29 through Day 36
Occurrence of solicited injection site reactogenicity events overall | Day 1 through Day 8
Occurrence of solicited injection site reactogenicity events overall | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 1 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 1 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 2 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 2 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 3 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 3 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 4 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 4 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 5 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 5 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events in Group 6 | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events in Group 6 | Day 29 through Day 36
Occurrence of solicited systemic reactogenicity events overall | Day 1 through Day 8
Occurrence of solicited systemic reactogenicity events overall | Day 29 through Day 36

SECONDARY OUTCOMES:
Comparison of geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 2 | Day 211
Comparison of geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 3 | Day 211
Comparison of geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 4 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 2 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 3 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 4 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 5 and Group 2 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 5 and Group 3 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 5 and Group 4 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 5 and Group 6 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 6 and Group 2 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 6 and Group 3 | Day 211
Comparison of geometric mean titer (GMT) (as measured by PRNT) to YF between Group 6 and Group 4 | Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 2 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 3 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 1 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 2 and Group 3 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 2 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN between Group 3 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 2 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 3 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 1 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 2 and Group 3 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 2 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR between Group 3 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 3 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 3 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 4 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 4 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 5 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 5 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 6 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 2 and Group 6 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 4 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 4 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 5 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 5 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 6 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 3 and Group 6 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 4 and Group 5 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 4 and Group 5 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 4 and Group 6 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 4 and Group 6 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 5 and Group 6 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination between Group 5 and Group 6 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 2 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 2 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 3 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 3 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 4 | Day 15 through Day 22
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF after vaccination with MVA-BN-YF in Group 6 compared to Group 4 | Day 36 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 2 and Group 3 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 2 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 2 and Group 5 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 2 and Group 6 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 3 and Group 4 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 3 and Group 5 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 3 and Group 6 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 4 and Group 5 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 4 and Group 6 | Day 1 through Day 211
Comparison of peak geometric mean titer (GMT) (as measured by PRNT) to YF between Group 5 and Group 6 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 1 through Day 211
Peak geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 1 through Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 15
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 22
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 36
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 43
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 50
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 1 | Day 57
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 15
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 22
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 36
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 43
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 50
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 2 | Day 57
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 15
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 22
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 36
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 43
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 50
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 3 | Day 57
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 15
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 22
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 36
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 43
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 50
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 4 | Day 57
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 15
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 211
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 22
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 36
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 43
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 50
Per-visit geometric mean titer (GMT) (as measured by ELISA) to MVA-BN in Group 6 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 1 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 2 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 3 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 4 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to VACV-WR in Group 6 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 2 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 3 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 4 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 5 | Day 57
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 15
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 211
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 22
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 36
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 43
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 50
Per-visit geometric mean titer (GMT) (as measured by PRNT) to YF in Group 6 | Day 57
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 1
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 15
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 211
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 22
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 29
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 36
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 43
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 50
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 1 | Day 57
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 1
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 15
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 211
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 22
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 29
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 36
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 43
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 50
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 2 | Day 57
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 1
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 15
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 211
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 22
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 29
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 36
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 43
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 50
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 3 | Day 57
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 1
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 15
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 211
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 22
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 29
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 36
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 43
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 50
Proportion of subjects seroconverting to MVA-BN (VACV-WR PRNT defined as PRNT50 = / > 2 and MVA-BN ELISA defined as titer = / > 50 or = / > 2-fold rise in ELISA antibody responses compared with baseline if baseline ELISA titer = / > 50) in Group 4 | Day 57
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 1
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 15
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 211
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 22
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 29
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 36
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 43
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 50
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 2 | Day 57
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 1
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 15
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 211
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 22
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 29
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 36
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 43
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 50
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 3 | Day 57
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 1
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 15
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 211
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 22
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 29
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 36
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 43
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 50
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 4 | Day 57
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 1
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 15
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 211
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 22
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 29
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 36
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 43
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 50
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 5 | Day 57
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 1
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 15
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 211
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 22
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 29
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 36
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 43
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 50
Proportion of subjects seroconverting to YF (defined as PRNT50 titer = / > 20 or = / > 4-fold increase in neutralizing antibody responses to YF compared with baseline if baseline PRNT50 titer = / > 20) in Group 6 | Day 57

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri